CLINICAL TRIAL: NCT03938883
Title: A Randomized Masked (Reading Center), Controlled, Prospective Pivotal Study of the Effectiveness and Safety of the EyeGate Ocular Bandage Gel, a 0.75% Crosslinked Hyaluronic Acid (HA) Applied Topically, Versus a Bandage Contact Lens (BCL) in Accelerating Re-epithelialization of Large Corneal Epithelial Defects in Patients Having Undergone Photorefractive Keratectomy (PRK).
Brief Title: Ocular Bandage Gel (OBG) Pivotal Trial in Patients Undergoing Photorefractive Keratectomy ("PRK")
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EYEGATE-034
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Ophthalmology; Photorefractive Keratectomy ("PRK"); Laser Assisted Surgery; Refractive Surgery
Keywords: Photorefractive Keratectomy, Corneal Defect

STUDY DESIGN:
Intervention Model Description: All subjects (all eyes) who receive any study treatment will be evaluable for safety analysis. All treatment assignments are assigned through 1:1 randomization with one eye designated as the "study eye" for statistical purposes. The final subject evaluability will be determined prior to breaking the code for masked treatment assignment and locking the database.
Who Masked: Outcomes Assessor
Masking Description: Masked images will be sent to a central reading center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Ocular Bandage Gel (OBG) (Experimental): Cross-linked Hyaluronic Acid 0.75%, regulated through CDRH (device). EyeGate Ocular Bandage Gel will be applied topically to both eyes (OU) four times a day. Ocular Bandage Gel use is discontinued once complete re-epithelialization has occurred in that eye.
  Interventions: Device: Ocular Bandage Gel (OBG)
- Bandage Contact Lens (BCL) (Other): standard-of-care post-operative intervention following PRK. BCL (Acuvue® Oasys plano lens) applied OU. Bandage contact lens use is discontinued once complete re-epithelialization has occurred in that eye.
  Interventions: Device: Bandage Contact Lens (BCL)

INTERVENTIONS:
Device: Ocular Bandage Gel (OBG) — A modified form of the natural polymer hyaluronic acid, which is a gel that possesses unique physical and chemical properties such as hydrating and healing when applied to the ocular surface. The ability of CMHA-S to adhere longer to the ocular surface, resist degradation and protect the ocular surface makes it well-suited for treating various ocular surface injuries including surgical trauma.
  Other Names: crosslinked thiolated carboxymethyl hyaluronic acid ("CMHA-S")
  Arms: Ocular Bandage Gel (OBG)
Device: Bandage Contact Lens (BCL) — A bandage contact lens protects an injured or diseased cornea from the mechanical rubbing of the blinking eyelids, therefore allowing it to heal. It is a normal (usually soft, but not always) contact lens has no power. It is not intended to improve your vision.
  Other Names: Acuvue Oasys
  Arms: Bandage Contact Lens (BCL)

SUMMARY:
Prospective, randomized, masked (reading center), controlled pivotal study of Ocular Bandage Gel (OBG) vs. a bandage contact lens (BCL) in subjects who have undergone bilateral photorefractive keratectomy (PRK).

DETAILED DESCRIPTION:
This is a prospective, randomized, masked (reading center), controlled pivotal study of Ocular Bandage Gel (OBG) vs. a Bandage Contact Lens (BCL) in subjects who have undergone bilateral photorefractive keratectomy (PRK).

Study subjects will be evaluated and, if eligible following PRK, will receive the study treatment in a 1:1 randomization with both eyes receiving the same treatment.

Sites will capture the time that PRK surgery OU is completed. Sites will enroll eligible subjects and randomly assign a subject to Treatment Group (OBG) or Control Group (BCL). One eye will be randomized as the designated "study eye" for statistical purposes.

The reading center will be masked as to the randomization assignments. Both eyes will receive the same randomized assignment and both eyes of each subject will be evaluated at all timepoints.

The defect in both eyes of all subjects will be measured starting at Day 2 (48 hours after PRK). The slit lamp photos are to be collected at 48 hours (±1 hour) from PRK completion in both eyes.

The BCL in the Control Group eyes will be removed daily starting at Day 2 for slit lamp photos. Slit lamp measurements, as well as photography of the epithelial defect (without and with fluorescein), will be taken of both eyes of all subjects. Photos will be evaluated by a masked reading center.

ELIGIBILITY:
Inclusion Criteria:

* Undergone PRK with a fresh epithelial defect.
* Best corrected visual acuity (BCVA) of 20/20 or better at baseline

Exclusion Criteria:

* History of systemic disorders that may affect post-operative healing.
* Corneal pathology that would affect wound re-epithelization.
* Use of medications that may affect the rate of corneal healing.
* Pregnant or lactating females.

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Complete corneal re-epithelialization on Day 3 | Day 3 (72 hours)
  Evaluated by a masked reading center using digital photography of fluorescein stained slit lamp photos and image analysis. Proportion of eyes following PRK surgery with complete corneal re-epithelization of the epithelial defect on Day 3 and no recurrent erosions.

SECONDARY OUTCOMES:
Time to corneal re-epithelialization | Day 3 (72 hours)
  Evaluated by a masked reading center using digital photography of fluorescein stained slit lamp photos and image analysis. Time to closure in eyes following PRK surgery with complete re-epithelialization and no recurrent erosions.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Wirostko, M.D., Study Director — EyeGate
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
No plan developed or decided upon at this time.

REFERENCES:
- [Background] Durrie DS, Wolsey D, Thompson V, Assang C, Mann B, Wirostko B. Ability of a new crosslinked polymer ocular bandage gel to accelerate reepithelialization after photorefractive keratectomy. J Cataract Refract Surg. 2018 Mar;44(3):369-375. doi: 10.1016/j.jcrs.2018.01.018. PMID 29703289